CLINICAL TRIAL: NCT03211858
Title: Six-month, Randomized, Open-label, Parallel-group Comparison of SAR341402 to NovoLog®/NovoRapid® in Adult Patients With Diabetes Mellitus Also Using Insulin Glargine, With a 6-month Safety Extension Period
Brief Title: Comparison of SAR341402 to NovoLog/NovoRapid in Adult Patients With Diabetes Mellitus Also Using Insulin Glargine
Acronym: GEMELLI1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC15081; 2017-000091-28 (EudraCT Number); U1111-1191-5775 (Other: UTN)
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2019-08-08 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus-Type 2 Diabetes Mellitus
MeSH Terms: interventions — Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR341402 (Experimental): SAR341402 subcutaneous (SC), before meals intake on top of once daily (QD) Insulin Glargine, up to Week 52.
  Interventions: Drug: Insulin aspart; Drug: Insulin glargine (HOE901)
- NovoLog/NovoRapid (Active Comparator): NovoLog/NovoRapid SC, before meals intake on top of QD Insulin Glargine, up to Week 52.
  Interventions: Drug: NovoLog/NovoRapid; Drug: Insulin glargine (HOE901)

INTERVENTIONS:
Drug: Insulin aspart — SAR341402 100 units per milliliters (U/mL) (dose range of 1 unit to 80 units) self-administered by SC injection, immediately (within 5-10 minutes) before meal intake. Dose adjusted to achieve a 2-hour postprandial plasma glucose (PPG <10 millimoles/liter [mmol/L] [<180 milligram/deciliter {mg/dL}]) while avoiding hypoglycemia.
  Arms: SAR341402
Drug: NovoLog/NovoRapid — NovoLog/NovoRapid 100 U/mL (dose range of 1 unit to 60 units) self-administered by SC injection, immediately (within 5-10 minutes) before meal intake. Dose adjusted to achieve a 2-hour postprandial plasma glucose (PPG <10 mmol/L [<180 mg/dL]) while avoiding hypoglycemia.
  Other Names: Insulin aspart
  Arms: NovoLog/NovoRapid
Drug: Insulin glargine (HOE901) — Insulin glargine 100 U/mL injected QD subcutaneously consistent with the local label. Doses adjusted to achieve glycemic target for fasting, preprandial plasma glucose between 4.4 to 7.2 mmol/L (80 to 130 mg/dL) without hypoglycemia.
  Other Names: Lantus

SUMMARY:
Primary Objective:

To demonstrate non-inferiority of SAR341402 versus NovoLog/NovoRapid in glycated hemoglobin A1c (HbA1c) change from baseline to Week 26 in participants with type 1 or type 2 diabetes mellitus (T1DM or T2DM) also using Lantus®.

Secondary Objectives:

* To assess the immunogenicity of SAR341402 and NovoLog/NovoRapid in terms of positive/negative status and anti-insulin antibody (AIA) titers during the course of the study.
* To assess the relationship of AIAs with efficacy and safety.
* To assess the efficacy of SAR341402 and NovoLog/NovoRapid in terms of proportion of participants reaching HbA1c lesser than (<) 7.0% and change in HbA1c, fasting plasma glucose (FPG), and self-measured plasma glucose (SMPG) profiles from baseline to Week 26 and Week 52 (only Week 52 for HbA1c).
* To assess safety of SAR341402 and NovoLog/NovoRapid.

DETAILED DESCRIPTION:
The study consisted of a 2-week screening period, a 26-week treatment period, a 26-week comparative safety extension period, and a 1-day follow-up period. The maximum study duration was 54 weeks per participant and a 1 day safety follow-up.

ELIGIBILITY:
Inclusion criteria :

* Participants with T1DM or T2DM (T2DM US only) diagnosed for at least 12 months, who have been treated with a multiple daily injection regimen with
* NovoLog/NovoRapid or insulin lispro (100 U/mL) in the last 6 months prior to screening visit AND
* insulin glargine (100 U/mL) in the last 6 months prior to screening visit OR insulin detemir (Levemir®) in the last 12 months prior to screening visit.

Exclusion criteria:

* At screening visit, age under legal age of adulthood.
* HbA1c <7.0% or greater than (>) 10% at screening.
* Less than 1 year on continuous insulin treatment.
* Use of insulin pump in the last 3 months before screening visit.
* Participants with incomplete baseline 7-point SMPG profile, defined as participants who do not have 7-point profiles with at least 5 points on at least 2 days in the week before randomization Visit 3.
* Participants with T1DM: Use of glucose lowering agents other than insulin including use of non-insulin injectable peptides in the last 3 months prior to screening.
* Participants with T2DM:

  * Use of glucagon-like peptide-1 (GLP-1) receptor agonists in the last 3 months before screening visit.
  * Use of oral antidiabetic drugs (OADs) not on stable dose in the last 3 months before screening visit (sulfonylureas was discontinued at baseline).
* At screening visit, body mass index (BMI) greater than or equal to (>=) 35 kilogram per meter square (kg/m^2) in participants with T1DM and >=40 kg/m^2 in participants with T2DM.
* Use of insulin other than:

  * insulin glargine 100 U/mL and NovoLog/NovoRapid or insulin lispro 100 U/mL as part of a multiple injection regimen in the last 6 months before screening visit, OR
  * insulin detemir 100 U/mL in the 12 months before screening visit and NovoLog/NovoRapid or insulin lispro 100 U/mL in the last 6 months before screening visit as part of a multiple injection regimen.
* Status post pancreatectomy.
* Status post pancreas and/or islet cell transplantation.
* Hospitalization for recurrent diabetic ketoacidosis in the last 3 months before screening visit.
* History of severe hypoglycemia requiring Emergency Room admission or hospitalization in the last 3 months before screening visit.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment or injectable drugs) during the study period.
* Pregnant or breastfeeding women.
* Women of childbearing potential not protected by highly effective method(s) of birth control.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2019-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (82):
- United States (42):
  - Investigational Site Number 8400040, Little Rock, Arkansas
  - Investigational Site Number 8400012, Concord, California
  - Investigational Site Number 8400002, Escondido, California
  - Investigational Site Number 8400030, Fresno, California
  - Investigational Site Number 8400004, Greenbrae, California
  - Investigational Site Number 8400014, La Jolla, California
  - Investigational Site Number 8400043, Los Angeles, California
  - Investigational Site Number 8400036, Pomona, California
  - Investigational Site Number 8400011, Santa Barbara, California
  - Investigational Site Number 8400013, Ventura, California
  - Investigational Site Number 8400037, Aurora, Colorado
  - Investigational Site Number 8400018, Englewood, Colorado
  - Investigational Site Number 8400031, New Port Richey, Florida
  - Investigational Site Number 8400027, Ocoee, Florida
  - Investigational Site Number 8400007, Atlanta, Georgia
  - Investigational Site Number 8400022, Columbus, Georgia
  - Investigational Site Number 8400032, Roswell, Georgia
  - Investigational Site Number 8400038, Arlington Heights, Illinois
  - Investigational Site Number 8400005, Des Moines, Iowa
  - Investigational Site Number 8400041, Metairie, Louisiana
  - Investigational Site Number 8400015, Rockville, Maryland
  - Investigational Site Number 8400042, Waltham, Massachusetts
  - Investigational Site Number 8400019, Flint, Michigan
  - Investigational Site Number 8400003, Omaha, Nebraska
  - Investigational Site Number 8400024, Henderson, Nevada
  - Investigational Site Number 8400028, New York, New York
  - Investigational Site Number 8400025, Morehead City, North Carolina
  - Investigational Site Number 8400010, Wilmington, North Carolina
  - Investigational Site Number 8400023, Fargo, North Dakota
  - Investigational Site Number 8400029, Bend, Oregon
  - Investigational Site Number 8400033, Chattanooga, Tennessee
  - Investigational Site Number 8400044, Austin, Texas
  - Investigational Site Number 8400009, Dallas, Texas
  - Investigational Site Number 8400035, Dallas, Texas
  - Investigational Site Number 8400021, Dallas, Texas
  - Investigational Site Number 8400017, Houston, Texas
  - Investigational Site Number 8400001, Houston, Texas
  - Investigational Site Number 8400020, Houston, Texas
  - Investigational Site Number 8400016, Mesquite, Texas
  - Investigational Site Number 8400034, Salt Lake City, Utah
  - Investigational Site Number 8400008, Renton, Washington
  - Investigational Site Number 8400039, Bridgeport, West Virginia
- Finland (4):
  - Investigational Site Number 2460006, Jyväskylä
  - Investigational Site Number 2460002, Kuopio
  - Investigational Site Number 2460004, Pori
  - Investigational Site Number 2460003, Seinäjoki
- Germany (5):
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760006, Essen
  - Investigational Site Number 2760004, Heidelberg
  - Investigational Site Number 2760005, Oldenburg in Holstein
  - Investigational Site Number 2760002, Pirna
- Hungary (10):
  - Investigational Site Number 3480012, Balatonfüred
  - Investigational Site Number 3480011, Budapest
  - Investigational Site Number 3480008, Budapest
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480005, Budapest
  - Investigational Site Number 3480004, Budapest
  - Investigational Site Number 3480007, Debrecen
  - Investigational Site Number 3480003, Nagykanizsa
  - Investigational Site Number 3480010, Nyíregyháza
  - Investigational Site Number 3480009, Szentendre
- Japan (10):
  - Investigational Site Number 3920009, Fukuyama-Shi
  - Investigational Site Number 3920008, Higashiosaka-Shi
  - Investigational Site Number 3920007, Kashiwara-Shi
  - Investigational Site Number 3920001, Koriyama-Shi
  - Investigational Site Number 3920005, Kumamoto
  - Investigational Site Number 3920003, Mito
  - Investigational Site Number 3920010, Osaka
  - Investigational Site Number 3920002, Sagamihara-Shi
  - Investigational Site Number 3920004, Shinjuku-Ku
  - Investigational Site Number 3920006, Ushiku-Shi
- Poland (7):
  - Investigational Site Number 6160004, Bialystok
  - Investigational Site Number 6160003, Krakow
  - Investigational Site Number 6160005, Krakow
  - Investigational Site Number 6160007, Lublin
  - Investigational Site Number 6160006, Nowy Sącz
  - Investigational Site Number 6160001, Poznan
  - Investigational Site Number 6160002, Warsaw
- Russia (4):
  - Investigational Site Number 6430001, Saint Petersburg
  - Investigational Site Number 6430002, Samara
  - Investigational Site Number 6430003, Saratov
  - Investigational Site Number 6430004, Tomsk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Garg SK, Wernicke-Panten K, Wardecki M, Kramer D, Delalande F, Franek E, Sadeharju K, Monchamp T, Mukherjee B, Shah VN. Efficacy and Safety of Insulin Aspart Biosimilar SAR341402 Versus Originator Insulin Aspart in People with Diabetes Treated for 26 Weeks with Multiple Daily Injections in Combination with Insulin Glargine: A Randomized Open-Label Trial (GEMELLI 1). Diabetes Technol Ther. 2020 Feb;22(2):85-95. doi: 10.1089/dia.2019.0382. PMID 31804851
- [Background] Garg SK, Wernicke-Panten K, Wardecki M, Kramer D, Delalande F, Franek E, Sadeharju K, Monchamp T, Miossec P, Mukherjee B, Shah VN. Safety, Immunogenicity, and Glycemic Control of Insulin Aspart Biosimilar SAR341402 Versus Originator Insulin Aspart in People with Diabetes Also Using Insulin Glargine: 12-Month Results from the GEMELLI 1 Trial. Diabetes Technol Ther. 2020 Jul;22(7):516-526. doi: 10.1089/dia.2020.0008. Epub 2020 Mar 31. PMID 32068436
- [Derived] Shah VN, Franek E, Wernicke-Panten K, Pierre S, Mukherjee B, Sadeharju K. Efficacy, Safety, and Immunogenicity of Insulin Aspart Biosimilar SAR341402 Compared with Originator Insulin Aspart in Adults with Diabetes (GEMELLI 1): A Subgroup Analysis by Prior Type of Mealtime Insulin. Diabetes Ther. 2021 Feb;12(2):557-568. doi: 10.1007/s13300-020-00992-x. Epub 2021 Jan 11. PMID 33432547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 82 centers in 7 countries. A total of 846 participants were screened between 02 August 2017 and 29 December 2017, of which 249 participants were screen failures. Screen failures were mainly due to glycated hemoglobin A1c (HbA1c) level lesser than (<) 7.0% or greater than (>) 10% at the screening visit.
Pre-assignment Details: Randomization was stratified by HbA1c at screening visit (<8%, greater than or equal to [>=] 8%), prior use of NovoLog/NovoRapid (Yes, No), geographical region (Europe, United States [US], Japan) and type 1 or 2 of diabetes mellitus (T1DM/T2DM [US only]). Assigned to arms in 1:1 ratio (SAR341402: NovoLog/NovoRapid).
Groups:
- SAR341402: SAR341402 100 units per milliliter (U/mL) subcutaneous (SC) injection, before meals intake on top of once daily (QD) Insulin Glargine, up to Week 52.
- NovoLog/NovoRapid: NovoLog/NovoRapid 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine,up to Week 52.
Period: Overall Study
Arm/Group | SAR341402 | NovoLog/NovoRapid
Started | 301 | 296
Treated | 301 | 296
Completed (Completed 12-month on treatment period.) | 264 | 263
Not Completed | 37 | 33
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 0 | 4
Not completed — Poor compliance to protocol | 6 | 2
Not completed — Non-serious Hypoglycemia | 1 | 0
Not completed — Other than specified above | 22 | 21

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- SAR341402: SAR341402 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- NovoLog/NovoRapid: NovoLog/NovoRapid 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- Total: Total of all reporting groups
Arm/Group | SAR341402 | NovoLog/NovoRapid | Total
Number analyzed (Participants) | 301 | 296 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (14.8) | 47.8 (15.4) | 48.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 119 | 241
  Male | 179 | 177 | 356
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, "Overall number of participants analyzed" = participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 300 | 293 | 593
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 37 | 37 | 74
    Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
    Black or African American | 11 | 8 | 19
    White | 248 | 242 | 490
    More than one race | 0 | 3 | 3
    Unknown or Not Reported | 1 | 1 | 2
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/meter square^2 (kg/m^2)] | 27.45 (4.58) | 27.46 (4.99) | 27.45 (4.78)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 19.5 (11.9) | 19.4 (11.8) | 19.5 (11.8)
Glycated Haemoglobin [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.00 (0.77) | 7.94 (0.70) | 7.97 (0.74)
Randomization Strata of Types of Diabetes [Count of Participants; unit: Participants]
  Type 1 Diabetes Mellitus | 250 | 247 | 497
  Type 2 Diabetes Mellitus | 51 | 49 | 100
Randomization Strata of Screening HbA1c Categories [Count of Participants; unit: Participants]
  HbA1c <8% | 143 | 138 | 281
  HbA1c >=8% | 158 | 158 | 316
Randomization Strata of Prior Use of NovoLog/NovoRapid [Count of Participants; unit: Participants] — Here, "No" signifies participant who had prior use of Humalog/Liprolog; "Yes" signifies prior use of NovoLog/NovoRapid.
  Participants
    No (Humalog/Liprolog) | 109 | 108 | 217
    Yes (NovoLog/NovoRapid) | 192 | 188 | 380
Randomization strata of geographical region [Count of Participants; unit: Participants]
  Europe | 98 | 99 | 197
  Japan | 33 | 32 | 65
  US | 170 | 165 | 335

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin A1c (HbA1c) From Baseline to Week 26
Description: All values up to Week 26 were taken into account in the analysis, regardless of adherence to treatment. Change in HbA1c was calculated by subtracting baseline value from Week 26 value. Missing changes at Week 26 were imputed using a retrieved dropout multiple imputation method (separately for participants who prematurely discontinued or completed treatment). Adjusted least square (LS) means and standard errors (SE) were obtained using an analysis of covariance (ANCOVA) model on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 26
Population: Analysis was performed on intent-to-treat (ITT) population, which included all randomized participants, irrespective of compliance with the study protocol and procedures.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
percentage of HbA1c | -0.38 (0.042) | -0.30 (0.041)
Statistical Analysis 1: Comparison: SAR341402 vs NovoLog/NovoRapid; Analysis was performed using ANCOVA with treatment group (SAR341402, NovoLog/NovoRapid), the randomization strata of geographical region, type of diabetes and prior use of NovoLog/NovoRapid as fixed categorical effects, as well as the continuous fixed covariate of baseline HbA1c value; Test type: Non-Inferiority — Non-inferiority of SAR341402 over NovoLog/NovoRapid was demonstrated if upper bound of the 2-sided 95% confidence interval (CI) of the difference between SAR341402 and NovoLog/NovoRapid was <0.3%. If non-inferiority was demonstrated, using a hierarchical step down testing procedure, the inverse non-inferiority of NovoLog/NovoRapid over SAR341402 was tested and was demonstrated if lower bound of the 2-sided 95% CI of the difference between SAR341402 and NovoLog/NovoRapid was > -0.3%; LS Mean difference = -0.08, 95% CI 2-sided [-0.192 to 0.039], Standard Error of Mean 0.059 — SAR341402 vs NovoLog/NovoRapid

2. Secondary Outcome: Change in HbA1c From Baseline to Week 52
Description: All values up to Week 52 were taken into account in the analysis, regardless of adherence to treatment. Change in HbA1c was calculated by subtracting baseline value from Week 52 value. Missing changes at Week 52 were imputed using a retrieved dropout multiple imputation method (separately for participants who prematurely discontinued or completed treatment). Adjusted LS means and SE were obtained using ANCOVA model on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
percentage of HbA1c | -0.25 (0.057) | -0.26 (0.059)

3. Secondary Outcome: Percentage of Participants With HbA1c <7% at Week 26 and Week 52
Description: Participants who had no available assessment at Week 26 and Week 52 were considered as non-responders.
Time Frame: Week 26 and Week 52
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
percentage of participants
  At Week 26 | 16.6 | 14.5
  At Week 52 | 19.6 | 18.2

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26 and Week 52
Description: All values up to Week 26 and Week 52 were taken into account in the analysis, regardless of adherence to treatment. Change in FPG at Week 26 and 52 was calculated by subtracting baseline value from Week 26 and Week 52 values, respectively. Missing changes at Week 26 and Week 52 were imputed using a retrieved dropout multiple imputation method (separately for participants who prematurely discontinued or completed treatment). Adjusted LS means and SE were obtained using ANCOVA analysis on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 26, and Week 52
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
millimoles per liter (mmol/L)
  At Week 26 | -0.49 (0.249) | -0.17 (0.245)
  At Week 52 | -0.10 (0.366) | -0.34 (0.359)

5. Secondary Outcome: Change in the Mean 24-hour Plasma Glucose Concentration From Baseline to Week 26 and Week 52
Description: Mean 24-hour plasma glucose concentration was calculated based on 7-point self-measured plasma glucose (SMPG) profiles with plasma glucose measurements before and 2-hours after each main meal and at bedtime. Mean 24-hour plasma glucose concentration was calculated for each profile and then averaged across profiles performed in the week before a visit. All calculated values up to Week 26 and Week 52 were taken into account in the analysis, regardless of adherence to treatment. Change in mean 24-hour plasma glucose concentration at Weeks 26 and 52 was calculated by subtracting baseline value from Week 26 and Week 52 values, respectively. Missing changes at Week 26 and Week 52 were imputed using a return-to-baseline multiple imputation method (values imputed as participant baseline plus an error). Adjusted LS means and SE were obtained using ANCOVA analysis on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 26, and Week 52
Population: Analysis was performed on ITT population. Here, "Overall number of participants analyzed" = participants with a baseline mean 24-hour plasma glucose concentration.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 295
mmol/L
  At Week 26 | -0.34 (0.120) | -0.53 (0.121)
  At Week 52 | 0.12 (0.144) | -0.18 (0.147)

6. Secondary Outcome: Change in Postprandial Plasma Glucose (PPG) Excursion From Baseline to Week 26 and Week 52
Description: Plasma glucose excursions were calculated at breakfast, lunch and dinner for each 7-point SMPG profile, as 2-hour PPG minus plasma glucose value obtained 30 minutes prior to start of the meal. Values of plasma glucose excursions at each visit were then calculated as the average across profiles performed in the week before the visit. All calculated values up to Week 26 and Week 52 were taken into account in the analysis, regardless of adherence to treatment. Change in PPG excursions at Weeks 26 and 52 was calculated by subtracting baseline value from Week 26 and Week 52 values, respectively. Missing changes at Week 26 and Week 52 were imputed using a return-to-baseline multiple imputation method (values imputed as participant baseline plus an error). Adjusted LS means and SE were obtained using ANCOVA analysis on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 26, and Week 52
Population: Analysis was performed on ITT population. Here, "Number analyzed" = participants with a baseline value for each specified category.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
mmol/L
  Week 26: At Breakfast: number analyzed (Participants) | 288 | 288
  Week 26: At Breakfast | 0.50 (0.232) | 0.65 (0.233)
  Week 26: At Lunch: number analyzed (Participants) | 290 | 291
  Week 26: At Lunch | 0.18 (0.230) | 0.12 (0.228)
  Week 26: At Dinner: number analyzed (Participants) | 290 | 292
  Week 26: At Dinner | 0.36 (0.243) | 0.66 (0.243)
  Week 52: At Breakfast: number analyzed (Participants) | 288 | 288
  Week 52: At Breakfast | 0.73 (0.253) | 0.91 (0.255)
  Week 52: At Lunch: number analyzed (Participants) | 290 | 291
  Week 52: At Lunch | 0.43 (0.252) | 0.34 (0.251)
  Week 52: At Dinner: number analyzed (Participants) | 290 | 292
  Week 52: At Dinner | 0.26 (0.255) | 0.51 (0.254)

7. Secondary Outcome: Change in 7-Point SMPG Profiles From Baseline to Week 26 and Week 52 Per Time Point
Description: 7-point SMPG profiles were measured at the following 7 points at each visit (Baseline, Week 26, and Week 52): before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, and bedtime. For each time point, the value at each visit was calculated as the average of values obtained for the same time point across profiles performed in the week before the visit.
Time Frame: Baseline, Week 26, and Week 52
Population: Analysis was performed on ITT population. Here, "Number analyzed" = participants with an available value at baseline, Week 26/Week 52 for the specified 7-point SMPG time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
mmol/L
  Week 26: Before Breakfast: number analyzed (Participants) | 254 | 253
  Week 26: Before Breakfast | -0.62 (4.48) | -0.50 (3.98)
  Week 26: 2 Hours After Breakfast: number analyzed (Participants) | 236 | 229
  Week 26: 2 Hours After Breakfast | -0.39 (4.97) | -0.30 (4.12)
  Week 26: Before Lunch: number analyzed (Participants) | 250 | 253
  Week 26: Before Lunch | -0.60 (4.14) | -0.60 (4.25)
  Week 26: 2 Hours After Lunch: number analyzed (Participants) | 246 | 251
  Week 26: 2 Hours After Lunch | -0.61 (4.54) | -0.62 (4.65)
  Week 26: Before Dinner: number analyzed (Participants) | 256 | 251
  Week 26: Before Dinner | -0.04 (4.87) | -0.78 (4.12)
  Week 26: 2 Hours After Dinner: number analyzed (Participants) | 240 | 245
  Week 26: 2 Hours After Dinner | -0.36 (4.71) | -0.25 (4.14)
  Week 26: Bedtime: number analyzed (Participants) | 239 | 238
  Week 26: Bedtime | -0.71 (5.13) | -0.54 (4.03)
  Week 52: Before Breakfast: number analyzed (Participants) | 240 | 229
  Week 52: Before Breakfast | -0.54 (4.80) | -0.31 (4.37)
  Week 52: 2 Hours After Breakfast: number analyzed (Participants) | 226 | 214
  Week 52: 2 Hours After Breakfast | -0.21 (4.30) | 0.05 (4.31)
  Week 52: Before Lunch: number analyzed (Participants) | 233 | 230
  Week 52: Before Lunch | 0.24 (4.64) | -0.13 (4.24)
  Week 52: 2 Hours After Lunch: number analyzed (Participants) | 231 | 227
  Week 52: 2 Hours After Lunch | 0.05 (5.01) | -0.37 (4.64)
  Week 52: Before Dinner: number analyzed (Participants) | 238 | 231
  Week 52: Before Dinner | 0.75 (5.59) | -0.06 (4.26)
  Week 52: 2 Hours After Dinner: number analyzed (Participants) | 227 | 227
  Week 52: 2 Hours After Dinner | 0.16 (4.60) | -0.17 (4.63)
  Week 52: Bedtime: number analyzed (Participants) | 220 | 215
  Week 52: Bedtime | -0.11 (4.98) | 0.10 (4.30)

8. Secondary Outcome: Number of Participants With at Least One Hypoglycemic Event
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because the participant was not capable of helping self. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=3.9 mmol/L (<=70 mg/dL) or plasma glucose level of <3.0 mmol/L (<54 mg/dL).
Time Frame: From first injection of investigational medicinal product (IMP) up to Week 26 or up to 1 day after last injection of IMP, whichever comes earlier, for Week 26 analysis, and from first injection of IMP up to 1 day after last injection of IMP for Week 52
Population: Analysis was performed on safety population that included all randomized participants who received at least one dose of IMP, analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
Participants
  Week 26: Any hypoglycemia | 291 | 285
  Week 26: Severe hypoglycemia | 12 | 10
  Week 26: Documented symptomatic <=3.9 mmol/L | 264 | 251
  Week 26: Documented symptomatic < 3.0 mmol/L | 207 | 193
  Week 52: Any hypoglycemia | 295 | 290
  Week 52: Severe hypoglycemia | 18 | 14
  Week 52: Documented symptomatic <=3.9 mmol/L | 274 | 267
  Week 52: Documented symptomatic hypo < 3.0 mmol/L | 223 | 220

9. Secondary Outcome: Number of Hypoglycemia Events Per Participant-Year
Description: Number of hypoglycemia events (any, severe and documented [both thresholds]) per participant-year of exposure were reported. Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because the participant was not capable of helping self. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=3.9 mmol/L (<=70 mg/dL) or plasma glucose level of <3.0 mmol/L (<54 mg/dL).
Time Frame: as for outcome 8
Population: Analysis was performed on safety population.
Measure: Number; unit: events per participant-year
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
events per participant-year
  Week 26: Any hypo | 73.33 | 69.71
  Week 26: Severe hypo | 0.14 | 0.10
  Week 26:Documented symptomatic hypo (<=3.9 mmol/L) | 40.36 | 36.37
  Week 26: Documented symptomatic hypo (<3.0 mmol/L) | 11.18 | 9.81
  Week 52: Any hypo | 66.00 | 64.46
  Week 52: Severe hypo | 0.12 | 0.08
  Week 52:Documented symptomatic hypo (<=3.9 mmol/L) | 35.68 | 33.73
  Week 52: Documented symptomatic hypo (<3.0 mmol/L) | 9.37 | 8.91

10. Secondary Outcome: Percentage of Participants With Hypersensitivity Reactions and Injection Site Reactions
Description: Participants with at least one treatment-emergent adverse event linked to hypersensitivity reaction and injection site reaction regardless of relationship to IMP during the main 6-month and the 12-month on-treatment periods was assessed and reported.
Time Frame: From first injection of IMP up to Week 26 or up to 1 day after last injection of IMP, whichever comes earlier, for Week 26 analysis, and from first injection of IMP up to 1 day after last injection of IMP for Week 52
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
percentage of participants
  Week 26: Hypersensitivity Reactions | 3.7 | 3.7
  Week 26: Injection site reactions | 0.7 | 1.4
  Week 52: Hypersensitivity Reactions | 5.6 | 7.1
  Week 52: Injection site reactions | 0.7 | 1.4

11. Secondary Outcome: Percentage of Participants With at Least One Positive Anti-Insulin Aspart Antibodies (AIA) Sample
Description: Participants with at least one positive AIA sample at baseline or at any time during the on-treatment period (Prevalence).
Time Frame: as for outcome 10
Population: Analysis was performed on AIA population, which included all participants who received at least one dose of IMP and had at least one AIA sample available for analysis during the on-treatment period, analyzed according to the treatment actually received. Here, "Number analyzed" = participants included in the AIA population at Week 26 and Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 298 | 292
percentage of participants
  At Week 26: number analyzed (Participants) | 296 | 292
  At Week 26 | 48.0 | 52.4
  At Week 52 | 54.7 | 58.2

12. Secondary Outcome: Percentage of Participants With Treatment-Induced, Treatment-Boosted and Treatment-Emergent Anti-insulin Aspart Antibodies (AIAs)
Description: AIA incidence were categorized as: treatment-induced, treatment-boosted AIAs, and treatment-emergent AIA. 1) Participants with treatment-induced AIAs were those who developed AIA following IMP administration (participants with at least one positive AIA sample at any time during on-treatment period, in those participants without pre-existing AIA or with missing baseline sample). 2) Participants with treatment-boosted AIAs were those with pre-existing AIAs that were boosted to a significant higher titer following IMP administration (participants with at least one AIA sample with at least a 4-fold increase in titers compared to baseline value at any time during on-treatment period). 3) Participants with treatment-emergent AIA were defined as participants with treatment-induced, or treatment-boosted AIAs.
Time Frame: as for outcome 10
Population: Analysis was performed on AIA population. Here, 'Number analyzed' = participants included in the AIA population at Week 26 and Week 52 and with negative or missing AIA status at baseline (for treatment-induced AIA) or with positive AIA status at baseline (for treatment-boosted AIA).
Measure: Number; unit: percentage of participants
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 298 | 292
percentage of participants
  Week 26: Treatment-Induced AIA: number analyzed (Participants) | 200 | 194
  Week 26: Treatment-Induced AIA | 23.0 | 28.4
  Week 26: Treatment-Boosted AIA: number analyzed (Participants) | 96 | 98
  Week 26: Treatment-Boosted AIA | 4.2 | 5.1
  Week 26: Treatment-Emergent AIA: number analyzed (Participants) | 296 | 292
  Week 26: Treatment-Emergent AIA | 16.9 | 20.5
  Week 52: Treatment-Induced AIA: number analyzed (Participants) | 202 | 194
  Week 52: Treatment-Induced AIA | 33.2 | 37.1
  Week 52: Treatment-Boosted AIA: number analyzed (Participants) | 96 | 98
  Week 52: Treatment-Boosted AIA | 9.4 | 13.3
  Week 52: Treatment-Emergent AIA | 25.5 | 29.1

13. Other Pre Specified Outcome: Change in Glycated Hemoglobin A1c From Baseline to Week 26 and Week 52: Subgroup Analysis by Prior Use of NovoLog/NovoRapid or Humalog/Liprolog
Description: All values up to Week 26 and Week 52 were taken into account in the analysis, regardless of adherence to treatment. Change in HbA1c at Week 26 and Week 52 was calculated by subtracting baseline value from Week 26 and Week 52 value, respectively. Missing changes at Week 26 and Week 52 were imputed using a retrieved dropout multiple imputation method (separately for participants who prematurely discontinued or completed treatment). Adjusted LS means and SE were obtained using ANCOVA model on data obtained from the multiple imputations (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 26 and Week 52
Population: Analysis was performed on ITT population and data was summarized separately for each treatment arm in each subgroup (based on the prior use of NovoLog/NovoRapid or Humalog/Liprolog).
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Prior NovoLog/NovoRapid Use: SAR341402: Participants with prior use of NovoLog/NovoRapid (as per randomization stratum), receiving SAR341402 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid: Participants with prior use of NovoLog/NovoRapid (as per randomization stratum), receiving NovoLog/NovoRapid 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- Prior Humalog/Liprolog Use: SAR341402: Participants with prior use of Humalog/Liprolog (as per randomization stratum), receiving SAR341402 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- Prior Humalog/Liprolog Use: NovoLog/NovoRapid: Participants with prior use of Humalog/Liprolog (as per randomization stratum), receiving NovoLog/NovoRapid 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
Arm/Group | Prior NovoLog/NovoRapid Use: SAR341402 | Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid | Prior Humalog/Liprolog Use: SAR341402 | Prior Humalog/Liprolog Use: NovoLog/NovoRapid
Number analyzed (Participants) | 192 | 188 | 109 | 108
percentage of HbA1c
  At Week 26 | -0.37 (0.052) | -0.33 (0.052) | -0.39 (0.070) | -0.24 (0.067)
  At Week 52 | -0.28 (0.065) | -0.26 (0.069) | -0.19 (0.091) | -0.26 (0.087)

14. Other Pre Specified Outcome: Number of Participants With at Least One Hypoglycemic Event: Subgroup Analysis by Prior Use of NovoLog/NovoRapid or Humalog/Liprolog
Description: as for outcome 8
Time Frame: as for outcome 10
Population: Analysis was performed on safety population and data was summarized separately for each treatment arm in each subgroup (based on the prior use of NovoLog/NovoRapid or Humalog/Liprolog).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior NovoLog/NovoRapid Use: SAR341402 | Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid | Prior Humalog/Liprolog Use: SAR341402 | Prior Humalog/Liprolog Use: NovoLog/NovoRapid
Number analyzed (Participants) | 192 | 188 | 109 | 108
Participants
  Week 26: Any hypoglycemia | 187 | 179 | 104 | 106
  Week 26: Severe hypoglycemia | 6 | 7 | 6 | 3
  Week 26: Documented symptomatic <=3.9 mmol/L | 170 | 162 | 94 | 89
  Week 26: Documented symptomatic < 3.0 mmol/L | 139 | 123 | 67 | 70
  Week 52: Any hypoglycemia | 190 | 184 | 105 | 106
  Week 52: Severe hypoglycemia | 10 | 9 | 8 | 5
  Week 52: Documented symptomatic <=3.9 mmol/L | 175 | 171 | 99 | 96
  Week 52: Documented symptomatic < 3.0 mmol/L | 149 | 138 | 74 | 82

15. Other Pre Specified Outcome: Number of Participants With Adverse Events: Subgroup Analysis by Prior Use of NovoLog/NovoRapid or Humalog/Liprolog
Description: Any untoward medical occurrence in a participant who received IMP was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during the main 6-month or 12-month on-treatment periods.
Time Frame: From first injection of IMP up to Week 26 or up to 1 day after last injection of IMP, whichever comes earlier for Week 26 analysis, and from first injection of IMP up to 1 day after last injection of IMP for Week 52
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Prior NovoLog/NovoRapid Use: SAR341402 | Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid | Prior Humalog/Liprolog Use: SAR341402 | Prior Humalog/Liprolog Use: NovoLog/NovoRapid
Number analyzed (Participants) | 192 | 188 | 109 | 108
Participants
  Week 26: Any TEAE | 92 | 94 | 64 | 52
  Week 52: Any TEAE | 115 | 109 | 69 | 59

16. Other Pre Specified Outcome: Percentage of Participants With Treatment-Induced, Treatment-Boosted and Treatment-Emergent Anti-insulin Aspart Antibodies (AIAs): Subgroup Analysis by Prior Use of NovoLog/NovoRapid or Humalog/Liprolog
Description: AIA incidence were categorized as: treatment-induced, treatment-boosted AIAs, and treatment-emergent AIA. 1) Participants with treatment-induced AIAs were those who developed AIA following IMP administration (participants with at least one positive AIA sample at any time during on-treatment period, in those participants without pre-existing AIA or with missing baseline sample. 2) Participants with treatment-boosted AIAs were those with pre-existing AIAs that were boosted to a significant higher titer following IMP administration (participants with at least one AIA sample with at least a 4-fold increase in titers compared to baseline value at any time during on-treatment period). 3) Participants with treatment-emergent AIA were defined as participants with treatment-induced, or treatment-boosted AIAs. Data was summarized separately for each treatment arm in each subgroup (based on the prior use of NovoLog/NovoRapid or Humalog/Liprolog).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Prior NovoLog/NovoRapid Use: SAR341402 | Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid | Prior Humalog/Liprolog Use: SAR341402 | Prior Humalog/Liprolog Use: NovoLog/NovoRapid
Number analyzed (Participants) | 191 | 185 | 107 | 107
percentage of participants
  Week 26: Treatment-Induced AIA: number analyzed (Participants) | 123 | 120 | 77 | 74
  Week 26: Treatment-Induced AIA | 18.7 | 28.3 | 29.9 | 28.4
  Week 26: Treatment-Boosted AIA: number analyzed (Participants) | 68 | 65 | 28 | 33
  Week 26: Treatment-Boosted AIA | 1.5 | 4.6 | 10.7 | 6.1
  Week 26: Treatment-Emergent AIA: number analyzed (Participants) | 191 | 185 | 105 | 107
  Week 26: Treatment-Emergent AIA | 12.6 | 20.0 | 24.8 | 21.5
  Week 52: Treatment-Induced AIA: number analyzed (Participants) | 123 | 120 | 79 | 74
  Week 52: Treatment-Induced AIA | 30.1 | 34.2 | 38.0 | 41.9
  Week 52: Treatment-Boosted AIA: number analyzed (Participants) | 68 | 65 | 28 | 33
  Week 52: Treatment-Boosted AIA | 5.9 | 15.4 | 17.9 | 9.1
  Week 52: Treatment-Emergent AIA | 21.5 | 27.6 | 32.7 | 31.8

17. Other Pre Specified Outcome: Change in Daily Insulin Dose From Baseline to Day 1, Week 26 and Week 52
Description: Change in daily insulin dose (basal, mealtime and total) was calculated by subtracting baseline value from Day1, Week 26 and Week 52 values respectively. Baseline was defined as the median of daily doses available in the week prior to the first injection of IMP (corresponding to doses of the pre-study insulin), value at Day 1 as the median of daily doses available in the week after the first injection of IMP (first doses of IMP), and value at Week 26 and Week 52 as the median of daily doses available in the week prior to each visit.
Time Frame: Baseline, Day 1, Week 26 and Week 52
Population: Analysis was performed on safety population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Units/kilogram (U/kg)
Arm/Group | SAR341402 | NovoLog/NovoRapid
Number analyzed (Participants) | 301 | 296
Units/kilogram (U/kg)
  Basal insulin dose at Day 1: number analyzed (Participants) | 290 | 283
  Basal insulin dose at Day 1 | -0.004 (0.036) | -0.000 (0.023)
  Mealtime insulin dose at Day 1: number analyzed (Participants) | 287 | 279
  Mealtime insulin dose at Day 1 | 0.003 (0.074) | 0.003 (0.091)
  Total insulin dose at Day 1: number analyzed (Participants) | 284 | 276
  Total insulin dose at Day 1 | -0.001 (0.076) | 0.002 (0.090)
  Basal insulin dose at Week 26: number analyzed (Participants) | 271 | 270
  Basal insulin dose at Week 26 | 0.005 (0.081) | 0.003 (0.088)
  Mealtime insulin dose at Week 26: number analyzed (Participants) | 268 | 265
  Mealtime insulin dose at Week 26 | -0.011 (0.133) | 0.011 (0.116)
  Total insulin dose at Week 26: number analyzed (Participants) | 263 | 262
  Total insulin dose at Week 26 | -0.007 (0.167) | 0.015 (0.170)
  Basal insulin dose at Week 52: number analyzed (Participants) | 253 | 253
  Basal insulin dose at Week 52 | 0.006 (0.085) | 0.005 (0.095)
  Mealtime insulin dose at Week 52: number analyzed (Participants) | 251 | 255
  Mealtime insulin dose at Week 52 | -0.001 (0.152) | 0.009 (0.123)
  Total insulin dose at Week 52: number analyzed (Participants) | 248 | 251
  Total insulin dose at Week 52 | 0.005 (0.175) | 0.013 (0.165)

18. Post Hoc Outcome: Change in Daily Insulin Dose From Baseline to Day 1, Week 26 and Week 52: Subgroup Analysis by Prior Use of NovoLog/NovoRapid or Humalog/Liprolog
Description: Change in daily insulin dose (basal, mealtime and total) was calculated by subtracting baseline value from Day 1, Week 26 and Week 52 values respectively. Baseline was defined as the median of daily doses available in the week prior to the first injection of IMP (corresponding to doses of the pre-study insulin), value at Day 1 as the median of daily doses available in the week after the first injection of IMP (first doses of IMP), and value at Week 26 and Week 52 as the median of daily doses available in the week prior to each visit.
Time Frame: Baseline, Day 1, Week 26, Week 52
Population: Analysis was performed on safety population and data was summarized separately for each treatment arm in each subgroup (based on the prior use of NovoLog/NovoRapid or Humalog/Liprolog). Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Prior NovoLog/NovoRapid Use: SAR341402 | Prior NovoLog/NovoRapid Use: NovoLog/NovoRapid | Prior Humalog/Liprolog Use: SAR341402 | Prior Humalog/Liprolog Use: NovoLog/NovoRapid
Number analyzed (Participants) | 192 | 188 | 109 | 108
U/kg
  Basal insulin dose at Day 1: number analyzed (Participants) | 182 | 182 | 108 | 101
  Basal insulin dose at Day 1 | -0.005 (0.037) | 0.0000 (0.021) | -0.002 (0.033) | -0.002 (0.026)
  Mealtime insulin dose at Day 1: number analyzed (Participants) | 183 | 179 | 104 | 100
  Mealtime insulin dose at Day 1 | -0.000 (0.073) | -0.003 (0.071) | 0.008 (0.075) | 0.013 (0.118)
  Total insulin dose at Day 1: number analyzed (Participants) | 180 | 178 | 104 | 98
  Total insulin dose at Day 1 | -0.006 (0.075) | -0.003 (0.077) | 0.006 (0.079) | 0.011 (0.111)
  Basal insulin dose at Week 26: number analyzed (Participants) | 174 | 173 | 97 | 97
  Basal insulin dose at Week 26 | 0.003 (0.087) | 0.009 (0.065) | 0.008 (0.070) | -0.006 (0.118)
  Mealtime insulin dose at Week 26: number analyzed (Participants) | 175 | 170 | 93 | 95
  Mealtime insulin dose at Week 26 | -0.009 (0.133) | 0.019 (0.114) | -0.015 (0.133) | -0.003 (0.121)
  Total insulin dose at Week 26: number analyzed (Participants) | 171 | 168 | 92 | 94
  Total insulin dose at Week 26 | -0.007 (0.171) | 0.027 (0.142) | -0.008 (0.159) | -0.006 (0.210)
  Basal insulin dose at Week 52: number analyzed (Participants) | 163 | 158 | 90 | 95
  Basal insulin dose at Week 52 | 0.004 (0.094) | 0.013 (0.088) | 0.010 (0.067) | -0.009 (0.105)
  Mealtime insulin dose at Week 52: number analyzed (Participants) | 164 | 160 | 87 | 95
  Mealtime insulin dose at Week 52 | -0.000 (0.156) | 0.015 (0.132) | -0.001 (0.147) | -0.001 (0.105)
  Total insulin dose at Week 52: number analyzed (Participants) | 161 | 157 | 87 | 94
  Total insulin dose at Week 52 | 0.003 (0.177) | 0.025 (0.169) | 0.009 (0.171) | -0.009 (0.156)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) weeks were collected from signature of the informed consent form up to the study completion (up to 52 Weeks) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment-emergent AEs, that is AEs that developed/worsened or became serious and deaths that occurred during the '12-month on-treatment period' (time from the first injection of IMP up to 1 day after the last injection of IMP). Analysis was performed on safety population.
Arm/Group | SAR341402 | NovoLog/NovoRapid
All-Cause Mortality (participants affected / at risk) | 1/301 | 2/296
Serious Adverse Events (participants affected / at risk) | 36/301 | 29/296
Other Adverse Events (participants affected / at risk) | 70/301 | 66/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR341402 (N=301) | NovoLog/NovoRapid (N=296)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Chronic Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (2)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 1 (1)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Biliary Dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis Chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 4 (9) | 2 (2)
Device Use Error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (9) | 2 (2)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prolymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycaemic Unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic Coma (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic Seizure (Nervous system disorders) | 3 (3) | 2 (4)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 10 (13) | 4 (5)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Intercapillary Glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR341402 (N=301) | NovoLog/NovoRapid (N=296)
Influenza (Infections and infestations) | 15 (15) | 12 (13)
Nasopharyngitis (Infections and infestations) | 34 (45) | 29 (39)
Upper Respiratory Tract Infection (Infections and infestations) | 22 (28) | 28 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT03211858/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT03211858/SAP_001.pdf